CLINICAL TRIAL: NCT02096367
Title: Immediate Effect of Cervical Posterior Muscles' and Gluteus Medius Muscle's Vibrations on Gait in Chronic Vascular Hemiplegia
Brief Title: Immediate Effect of Postural Muscle's Vibrations on Gait in Chronic Vascular Hemiplegia
Acronym: VIBR-AVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: École Normale Supérieure de Cachan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIBR-AVC
Record Dates: First submitted 2014-03-12; First posted 2014-03-26 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Hemiplegia; Stroke
Keywords: vibrations; stroke; posture; gait; readaptation
MeSH Terms: conditions — Hemiplegia; Stroke | interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemiplegia after vascular stroke (Experimental): * Muscle vibration stimulation
  * Gait analysis with Gait Rite : quantitative and spatio-temporal gait parameters
  * Kinematic gait analysis in lower limb measured by optoelectronic system (Optitrack).
  * Analysis of static posture on force platform
  * Evaluation of the gait on treadmill during 2 minutes
  Interventions: Other: Gait analysis; Other: Kinematic gait analysis in lower limb; Other: Analysis of static posture; Other: Gait on treadmill; Device: Muscle vibration stimulation

INTERVENTIONS:
Other: Gait analysis
  Other Names: Gait analysis system : Gait Rite®
Other: Kinematic gait analysis in lower limb
  Other Names: Optoelectronic system : Optitrack
Other: Analysis of static posture
  Other Names: Force platform Feetest® (Technoconcept, France)
Other: Gait on treadmill — Treadmill during 2 minutes
Device: Muscle vibration stimulation — Vibration stimulation at a 70 Hz frequency of biceps brachii muscle (sham), posterior neck muscles and gluteus medius muscle on the hemiplegic side
  Other Names: Device : VB 115 Vibrasens© (Technoconcept, France)

SUMMARY:
Balance disorders are very common after strokes and often last for long periods of time. Their origin is multifactorial and their impact on the daily lives of patients are particularly important, especially on gait.

The vibration technology for rehabilitation was already studied in static posture with force plats but their impact on gait have yet to be evaluated.

This present study aims at investigating the effects of vibrations applied by an approved medical device to the posterior neck muscles and the gluteus medius - major actors of proprioception and posture mechanisms - on gait disorders in patients with hemiplegia during the chronic phase after stroke.

DETAILED DESCRIPTION:
An inclusion medical exam will occur in order to explain the protocol to the patients, to receive their written informed consent and to check the inclusion and absence of non-inclusion criteria.

The study visit will happen in a 2 weeks' time span at most after the inclusion exam.

During the study visit, the patients will undergo:

* A quantitative gait analysis with Gait Rite and Optitrack before any intervention;
* Then, in a randomized order:

  * A vibration stimulation on a non-postural muscle (biceps brachii muscle) in order to get a control stimulation (or "sham") with a new gait analysis with Gait Rite and Optitrack during the stimulation, then 2 and 10 minutes after it stopped,
  * A vibration stimulation of the posterior neck muscles on the hemiplegic side, with a new gait analysis with Gait Rite and Optitrack during the stimulation, then 2 and 10 minutes after it stopped. The precise stimulation location will be located by the pressures centre deviation on a medio-lateral axis on a strength platform (this area can vary for a few centimetres from patient to patient),
  * In order to assess the secondary outcome aiming at defining the best stimulation location, a vibration stimulation of the gluteus medius on the hemiplegic side, with a new gait analysis with Gait Rite and Optitrack during the stimulation, then 2 and 10 minutes after it stopped. In the same way than for the neck muscles, the scouting of the precise location will be assessed facing the greater trochanter by the pressures centre deviation on a medio-lateral axis on a strength platform.

The realisation of the entire protocol will last approximately 90 minutes.

At the end of the test, an optoelectronic recording by Optitrack will be realised on a treadmill in order to highlight potential differences between the gait on the ground and trained gait at comfortable speed for 2 minutes maximum.

ELIGIBILITY:
Inclusion Criteria:

Hemiplegic subjects after stroke:

* Men or women aged over 18
* Stroke due to ischemic or haemorrhagic cause
* More than 6 months after stroke
* First episode of stroke
* Gait asymmetry before stimulation
* Able to walk more than 100 meters with or without cane
* Written informed consent

Exclusion Criteria:

* Orthopaedic or rheumatologic disorders impeding the good realisation of the measurement
* Adults under legal protective regimen or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of monopodal stance on the hemiplegic side | Day 0
  Improvement of the percentage of monopodal stance on the hemiplegic side during walking after stimulation by vibrations measured by quantitative gait analysis with Gait Rite

SECONDARY OUTCOMES:
Spatio-temporal gait parameters | Day 0
  Spatio-temporal gait parameters : speed, step time, time of double stance, time of swing, length and width of step
Kinematic gait parameters in lower limb | Day 0
  Kinematic gait parameters in lower limb (hip, knee, ankle) measured by optoelectronic system (Optitrack).
Static posture asymmetry | Day 0
  Analysis of static posture on force platform
Gait parameters on treadmill | Day 0
  Evaluation of gait parameters during 2 minutes on treadmill, measured by optoelectronic system (Optitrack).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Bonan, MD, PhD, Principal Investigator — CHU Rennes - Service de Médecine Physique et de Réadaptation
Locations (1):
- CHU Rennes - Pontchaillou Hospital, Rennes, Brittany Region, France